CLINICAL TRIAL: NCT05837793
Title: Evaluation of Postoperative Outcomes of Minimally Invasive Distal Pancreatectomy for Left-sided Pancreatic Tumors Based on the Modified Frailty Index: A Retrospective Cohort Study
Brief Title: Modified Frailty Index for Minimally Invasive Distal Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Song Cheol Kim (Other)
Responsible Party: Sponsor-Investigator, Song Cheol Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: 2022-1709
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- frail: The mFi categorizes patients with a score of 0.27 or higher as frail and those with a score below that as the non-frail group.
  Interventions: Behavioral: Modified frailty index
- and non-frail: The mFi categorizes patients with a score of 0.27 or higher as frail and those with a score below that as the non-frail group.
  Interventions: Behavioral: Modified frailty index

INTERVENTIONS:
Behavioral: Modified frailty index — The mFI includes the following 11 items from the National Surgical Quality Improvement Program (NSQIP): diabetes; functional status (not independent); chronic obstructive pulmonary disease (COPD) or pneumonia; congestive heart failure; history of myocardial infarction; hypertension requiring medication; peripheral vascular disease or rest pain; impaired sensorium; history of either transient ischemic attack or cerebrovascular accident; history of cerebrovascular accident with neurologic deficit; and prior percutaneous coronary intervention, previous coronary surgery, or history of angina.

SUMMARY:
This study aims to investigate the difference in postoperative complications according to the modified Frailty Index (mFI) in patients who underwent minimally invasive distal pancreatectomy for pancreatic tumors at the Asan Medical Center's Department of Hepato-Biliary-Pancreatic Surgery from 2005 to 2019. It also seeks to confirm the utility of mFI as a predictive factor for postoperative complications in frail patients in the future.

DETAILED DESCRIPTION:
Distal pancreatectomy is a surgery performed to treat tumors in the distal pancreas. The minimally invasive approach to this surgery has become the standard due to its shorter hospital stay, quicker recovery, less pain, and similar complication rates compared to open surgery, especially for benign tumors. In selected patients with malignant tumors, minimally invasive distal pancreatectomy has gradually expanded to a state where it is not inferior to open surgery in terms of postoperative complications and long-term prognosis. As the average lifespan increases, elderly patients with comorbidities are steadily increasing in numbers among those who undergo distal pancreatectomy. However, predicting postoperative complications and mortality rates for these patients is still difficult. Simple yet effective predictive factors for postoperative complications are needed. The Canadian Study of Health and Aging has created a standardized frailty index (CSHA-FI) as a tool for predicting frailty in elderly patients, and a modified Frailty Index (mFI) has been developed for easy use. The mFI has been reported as a predictor of postoperative morbidity and mortality rates after colorectal and vascular surgery. This study aims to investigate whether mFI can be used as a predictive factor for postoperative morbidity and mortality rates in patients who undergo minimally invasive distal pancreatectomy and to utilize it for clinical treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of patients who underwent minimally invasive distal pancreatectomy for pancreatic body or tail tumors between January 2005 and December 2019.

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to investigate the trend of frailty among patients who underwent minimally invasive pancreaticoduodenectomy for pancreatic head tumors between January 2005 and December 2019, using data collected until October 31, 2022. Based on an estimated 150 surgeries per year, the sample size is expected to be around 2000 patients. Frailty will be defined as mFI of 0.27 or higher, with an estimated prevalence of 3% among this patient population. The study will analyze the differences and severity of postoperative complications between frail and non-frail patients, while also examining the trend of frailty over the 15-year period. The expected sample size for the study is around 2000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Postoperative outcomes | 6 months
  Comparison of the Postoperative outcomes according to the mFI

CONTACTS AND LOCATIONS:
Overall Officials: Song Cheol Kim, MD. PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park Y, Hwang DW, Lee JH, Song KB, Jun E, Lee W, Kwak BJ, Kim SC. Evaluation of postoperative outcomes of minimally invasive distal pancreatectomy for left-sided pancreatic tumors based on the modified frailty index: a retrospective cohort study. Int J Surg. 2023 Nov 1;109(11):3497-3505. doi: 10.1097/JS9.0000000000000670. PMID 37598358